CLINICAL TRIAL: NCT03011320
Title: An Exploratory, Open-label Study of the Folic Acid-tubulysin Conjugate EC1456 in Ovarian Cancer Subjects Undergoing Cytoreductive Surgery
Brief Title: An Exploratory Study of the Folic Acid-tubulysin Conjugate EC1456 in Ovarian Cancer Subjects Undergoing Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Endocyte (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EC1456-02
Record Dates: First submitted 2016-12-19; First posted 2017-01-05 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Ovary Cancer
Keywords: ovarian cancer; specimen collection
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Folic Acid; Leucovorin; technetium 99m etarfolatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): Injection of unlabeled etarfolatide followed by etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection, followed by a single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT) scan.
  One dose of 4 mg/m2 EC1456 at <8 hours prior to surgery
  Interventions: Drug: EC1456; Drug: 99mTc-Etarfolatide
- Cohort 2 (Experimental): Injection of unlabeled etarfolatide followed by etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection, followed by a single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT) scan.
  One dose of 4 mg/m2 EC1456 at 48±4 hours prior to surgery
  Interventions: Drug: EC1456; Drug: 99mTc-Etarfolatide
- Cohort 3 (Experimental): Injection of unlabeled etarfolatide followed by etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection, followed by a single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT) scan.
  One dose of 8 mg/m2 EC1456 at <8 hours prior to surgery
  Interventions: Drug: EC1456; Drug: 99mTc-Etarfolatide
- Cohort 4 (Experimental): Injection of unlabeled etarfolatide followed by etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection, followed by a single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT) scan.
  One dose of 8 mg/m2 EC1456 at 48±4 hours prior to surgery
  Interventions: Drug: EC1456; Drug: 99mTc-Etarfolatide

INTERVENTIONS:
Drug: EC1456 — intravenous (IV) bolus dose
  Other Names: folate (vitamin B-9) and tubulysin B hydrazide small molecule conjugate
Drug: 99mTc-Etarfolatide — Injection of unlabeled etarfolatide followed by etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection, followed by a single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT) scan.
  Other Names: EC20; etarfolatide

SUMMARY:
This study looks to enroll subjects with ovarian cancer who will be having standard of care surgery to remove ovarian cancer tumors. The main aim of this study is to be able to observe how EC1456 has been taken in and broken down inside tumors. The effect of EC1456 on the tumor will also be studied. This study will also help us compare the amount of EC1456 seen in tumors and how the tumors are imaged by the 99mTc-etarfolatide single-photon emission tomography (SPECT) or single-photon emission tomography with in-line x-ray computed tomography (SPECT/CT).

All subjects will undergo a 99mTc-etarfolatide SPECT or SPECT/CT scan within 2 weeks prior to EC1456 administration.

Individual subjects will then receive 1 of the following 2 doses of EC1456 pre-operatively:

* 4 mg/m2
* 8 mg/m2

EC1456 will be administered at 1 of the following 2 time points:

* <8 hours before planned surgery
* 48±4 hours before planned surgery

Blood will be collected for pharmacokinetic (PK) studies right after EC1456 dosing and again right before surgery. At the time of surgery, tumor samples will be removed and sent to Endocyte for analysis.

DETAILED DESCRIPTION:
Study EC1456-02 is an exploratory, open-label study that seeks to enroll subjects with ovarian cancer who will be undergoing therapeutic debulking surgery.

All subjects will undergo a 99mTc-etarfolatide scan within 2 weeks prior to EC1456 administration. Briefly, prior to the 99mTc-etarfolatide imaging procedure, all subjects will receive one intravenous (IV) injection of folic acid or unlabeled etarfolatide, followed within 1 to 3 minutes by an injection of 99m Tc-etarfolatide (i.e., etarfolatide labeled with 740 to 925 megabecquerels (MBq) [20 to 25 millicuries (mCi)] of sodium pertechnetate Tc-99m injection).

Individual subjects will receive 1 of the following 2 doses of EC1456 pre-operatively:

* 4 milligrams (mg)/meter (m)2
* 8 milligrams (mg)/meter (m)2

EC1456 will be administered at 1 of the following 2 time points:

* <8 hours before planned surgery
* 48±4 hours before planned surgery

The 4 mg/m2 dose of EC1456 administered <8 hours prior to surgery will be the first dose cohort to enroll. Once enrollment to this cohort is complete, the remaining cohorts will be open for enrollment. Assignment to specific cohorts will be determined by the Sponsor based on data assessed from previously enrolled subjects. Two to six subjects will be enrolled per cohort as shown below.

* Cohort 1: 4 mg/m2 EC1456 <8 hours prior to surgery
* Cohort 2: 4 mg/m2 EC1456 48±4 hours prior to surgery
* Cohort 3: 8 mg/m2 EC1456 <8 hours prior to surgery
* Cohort 4: 8 mg/m2 EC1456 48±4 hours prior to surgery

In the event of unexpected results, lower, intermediate or higher EC1456 levels up to 12.5 mg/m2, the highest determined safe dose of EC1456 as defined by the parallel phase I study EC1456-01, may be explored.

The first on-study procedure will be SPECT or SPECT/CT with 99mTc-etarfolatide. SPECT or SPECT/CT scans will be acquired within 2 weeks prior to EC1456 administration as specified in the Imaging Operations Manual.

EC1456 will be administered pre-operatively as an intravenous (IV) bolus infusion at 1 of 2 time points:

1. < 8 hours preceding surgery or
2. 48±4 hours preceding surgery.

At 2 time points:

1. within approximately 15 (±5) minutes post-EC1456 administration and
2. at the start of surgery, approximately 5 mL of whole blood will be drawn for EC1456 analyses.

Tissues to be collected at surgery, if present, include: sample of 1 or both ovaries, endometrium, omentum, ascitic fluid and/or selected lesions as identified by the surgeon or sponsor. The location of each sample will be annotated such that the ex vivo analysis may be correlated with the SPECT/CT image post-surgery. Samples of tumor tissue will be collected at the time of surgery, aliquoted into collection vials, and placed on dry ice or in buffered formalin.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand, and have signed an approved informed consent form (ICF).
2. Subjects must have cytologically or pathologically confirmed advanced ovarian cancer and be scheduled for primary, interval, or secondary, cytoreductive surgery as a part of standard of care for treatment of ovarian cancer, and have at least 1 lesion that can be removed at surgery.
3. Subject must be ≥18 years of age.
4. Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
5. Subjects with central nervous system (CNS) metastases must be neurologically stable and off of steroids for at least 14 days before pre-registration. Subjects with asymptomatic CNS metastatic disease without associated edema, shift, and a requirement for steroids or anti-seizure medications may be eligible after discussion with the sponsor's medical monitor.
6. Subjects must have recovered (to baseline/ stabilization) from prior chemo- or radiotherapy and associated acute toxicities must have resolved to a NCI CTCAE v4 Grade 1 or less, with the exception of alopecia.
7. Subject must have adequate organ function:

   * Bone marrow reserve:

     * Absolute neutrophil count ≥1.5 × 109/L.
     * Platelets ≥100 × 109/L.
     * Hemoglobin ≥9 g/dL.
   * Cardiac:

     * Left ventricular ejection fraction (LVEF) ≥ the institutional lower limit of normal. LVEF must be evaluated within 28 days prior to the dose of EC1456.
     * Cardiac Troponin I within normal limits.
     * Electrocardiogram QT segment corrected by the method of Fridericia QTcFridericia (QTcF) < 450 msec on at least 2 of 3 screening ECG's. On site determination of QTcF may be used for screening purposes.
   * Hepatic:

     * Total bilirubin ≤1.5 × the upper limit of normal (ULN).
     * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST

       * 3.0 × ULN, or ≤5.0 × ULN for subjects with liver metastases.
     * Renal: Serum creatinine ≤1.5 × ULN, or for subjects with serum creatinine >1.5 × ULN, creatinine clearance ≥50 mL/min.
8. Subjects of childbearing potential:

   * All women of childbearing potential MUST have a negative urine or serum pregnancy test within 1 week prior to the 99mTc-etarfolatide imaging procedure and within 1 week prior to the dose of EC1456.
   * Women of childbearing potential must practice an effective method of birth control (e.g., oral, transdermal or injectable contraceptives, intrauterine device [IUD], or double-barrier contraception, such as diaphragm and spermicidal jelly) for the duration of their participation in

Exclusion Criteria:

1. In the opinion of the investigator, a subject's physical condition might create a hardship for tolerating the radionuclide imaging procedures or a single administration of EC1456 (e.g., due to pain or dyspnea in prolonged supine positions).
2. Use of the following medications within 6 months prior to EC1456 administration: amiodarone, disopyramide, dofetilide, dronedarone, flecanamide, ibutilide, quinidine, or sotalol.
3. Subject has a co-morbid medical condition that, in the opinion of the investigator, is known to have a major impact on the pharmacokinetics (PK), distribution, metabolism, or elimination of either small molecule drug conjugate (SMDC).
4. Subject has known active hepatitis B or hepatitis C.
5. Subject has active uncontrolled infection(s).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
To assess tumor penetration of EC1456 in frozen tissue | 18 months
  Measure and characterize intratumoral levels of EC1456, and metabolites, by liquid chromatography-tandem mass spectrometry (LC-MS/MS). All results will be descriptive and exploratory.

SECONDARY OUTCOMES:
To assess tumor penetration EC1456 in formalin fixed tissue samples (intratumoral levels of EC1456 in tissue blocks using anti-tubulysin IHC testing) | 18 months
  Measurement and characterization of intratumoral levels of EC1456 in the tissue blocks and assess if there is detectable penetration of the drug into the tumor using anti-tubulysin immunohistochemistry (IHC) testing. All results will be descriptive and exploratory.
To assess correlation of tumor penetration of EC1456 with tumor uptake of 99m-Tc etarfolatide in SPECT or SPECT/CT scan | 18 month
  Using the measures of tumor penetration, see if the SPECT or SPECT/CT scan correlates with etarfolatide update in the 99m-TC etarfolatide SPECT or SPECT/CT scans. All results will be descriptive and exploratory.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Armour, MB ChB, BSc, MSc, MD, MRCP, Study Director — Endocyte
Locations (2):
- Levine Cancer Institute-Concord/Clinical Trials, Concord, North Carolina, United States
- Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No